CLINICAL TRIAL: NCT03208244
Title: Pan-genotypic Direct Acting Antiviral Therapy in Donor HCV-positive to Recipient HCV-negative Heart Transplant
Brief Title: DAA Treatment in Donor HCV-positive to Recipient HCV-negative Heart Transplant
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Protocol transitioned to standard of care, no funding available to support research work
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Raymond Chung, Director of Hepatology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017P001427
Record Dates: First submitted 2017-07-03; First posted 2017-07-05 (Actual); Results first posted 2022-06-02 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: End Stage Heart Disease; Hepatitis C
Keywords: Heart Disease; Heart Transplant; HCV; Hepatitis C
MeSH Terms: conditions — Hepatitis C; Heart Diseases

STUDY DESIGN:
Intervention Model Description: Received heart transplant from HCV+ donor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with Direct Acting Antiviral for HCV (Experimental): 12 weeks of treatment with HCV Direct Acting Antiviral tablet
  Interventions: Drug: Clinically prescribed direct acting antiviral

INTERVENTIONS:
Drug: Clinically prescribed direct acting antiviral — HCV treatment for 12 weeks
  Other Names: DAA treatment

SUMMARY:
This is a proof of concept, single center study for the donation of HCV-positive hearts to HCV negative recipient patients, with preemptive, interventional treatment with 12 weeks of commercially available DAA therapy to prevent HCV transmission upon transplantation.

DETAILED DESCRIPTION:
The goal of this study is to determine if preoperative dosing and sustained administration of pan-genotypic DAA therapy after cardiac transplantation prevents the transmission of hepatitis C virus (HCV) infection from an HCV-positive donor heart to an HCV naïve recipient.

ELIGIBILITY:
Inclusion Criteria:

* Recipient is Age ≥ 18 years
* Serum ALT within normal limits with no history of liver disease
* Lack of sensitization (i.e. PRA < 20%) that would be expected to result in a high likelihood of needing aggressive immunosuppression to treat rejection

Exclusion Criteria:

* Sensitization (i.e. PRA >20%)
* Any liver disease in recipient
* Albumin < 3g/dl or platelet count < 75 x 103/mL
* Need for dual organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond L Chung, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Masschusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Anticipate to share coded data with collaborators
Supporting Information: Study Protocol
Time Frame: Anticipate data would be available to share within 6 months after the final patient completes the study.
Access Criteria: Coded data would be shared with collaborators who have received IRB approval to use the data and have been approved by the PI for their collaboration.

REFERENCES:
- [Derived] Bethea ED, Gaj K, Gustafson JL, Axtell A, Lebeis T, Schoenike M, Turvey K, Coglianese E, Thomas S, Newton-Cheh C, Ibrahim N, Carlson W, Ho JE, Shah R, Nayor M, Gift T, Shao S, Dugal A, Markmann J, Elias N, Yeh H, Andersson K, Pratt D, Bhan I, Safa K, Fishman J, Kotton C, Myoung P, Villavicencio MA, D'Alessandro D, Chung RT, Lewis GD. Pre-emptive pangenotypic direct acting antiviral therapy in donor HCV-positive to recipient HCV-negative heart transplantation: an open-label study. Lancet Gastroenterol Hepatol. 2019 Oct;4(10):771-780. doi: 10.1016/S2468-1253(19)30240-7. Epub 2019 Jul 26. PMID 31353243

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between 11/2017 and 4/1/2021
Pre-assignment Details: 7 participants received transplant with an HCV NAT negative organ and did not meet protocol criteria for DAA treatment.
Period: Overall Study
Arm/Group | Treatment With Direct Acting Antiviral for HCV
Started | 33
Completed | 32
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Number of subjects initiating treatment with DAA
Arm/Group | Treatment With Direct Acting Antiviral for HCV
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants] — Sex at birth as documented in the medical record.
  Participants
    Female | 10
    Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 28
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Undetectable HCV RNA at 12 Weeks Post Treatment
Description: Negative HCV viral RNA at 12 weeks after the last dose of treatment.
Time Frame: 12 weeks post treatment
Population: number of subjects active on study at 12 weeks post DAA treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Direct Acting Antiviral for HCV
Number analyzed (Participants) | 30
Participants | 30

2. Secondary Outcome: Number of Participants With Adverse Events and Clinically Significant Out of Range Lab Values of DAA Therapy in Patients Undergoing Cardiac Transplantation
Description: Safety and tolerablity of commercially available DAA therapy in the cardiac transplant patient will be monitored by quantifying the number of treatment related adverse events per patient and evaluating out of range laboratory results as compared to baseline/pretreatment values per patient.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Direct Acting Antiviral for HCV
Number analyzed (Participants) | 33
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the dosing period from date of first dose through date of last dose, an average of 12 weeks.
Description: Adverse events were consider if related or possibly related to DAA treatment or receipt of an HCV viremic organ. Expected side effects and/or complications related to clinical transplantation were not captured or assessed.
Arm/Group | Treatment With Direct Acting Antiviral for HCV
All-Cause Mortality (participants affected / at risk) | 1/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

LIMITATIONS AND CAVEATS:
Protocol was terminated prior to completion, primarily due to lack of resources (research staffing and funding) and clinical team moving HCV+ donor to HCV- recipient transplants to standard of care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/44/NCT03208244/Prot_SAP_000.pdf